CLINICAL TRIAL: NCT06785909
Title: The Role of Proprioceptive, Fear-related and Inflammatory Factors in the Persistence of Pregnancy-related Lumbopelvic Pain in Pregnant Women.
Brief Title: Proprioceptive, Fear-related and Inflammatory Factors in the Persistence of Pregnancy-related Lumbopelvic Pain.
Acronym: PROFit
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Collaborators: KU Leuven (Other)
Responsible Party: Principal Investigator, Lotte Janssens, Prof. dr., Hasselt University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: S69463
Record Dates: First submitted 2025-01-13; First posted 2025-01-21 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Low Back Pain; Lumbopelvic Pain; Pelvic Girdle Pain
Keywords: postural control; body perception; psychological factors; inflammation
MeSH Terms: conditions — Low Back Pain; Pelvic Girdle Pain; Inflammation | interventions — Psychology

STUDY DESIGN:
Intervention Model Description: Pregnant women without PLPP at the time of inclusion are followed from the first pregnancy trimester until 9 months postpartum. Assessments are performed during the first and third trimester, and 6 weeks and 9 months postpartum.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Primiparous pregnant women (Other): Pregnant women without PLPP at the time of inclusion are followed from the first pregnancy trimester until 9 months postpartum. Assessments are performed during the first and third trimester, and 6 weeks and 9 months postpartum.
  Interventions: Behavioral: Assessment of postural control, body perception, psychosocial factors and inflammation

INTERVENTIONS:
Behavioral: Assessment of postural control, body perception, psychosocial factors and inflammation — Behavioral assessment of postural control, lumbar proprioceptive use during postural control, back-specific body perception, psychosocial factors (incl. fear of movement, pain catastrophizing, sense of coherence, fear-avoidance beliefs, (pregnancy-related) depression, anxiety and stress) and inflammatory mediators.

SUMMARY:
Pregnancy-related lumbopelvic pain (PLPP) affects 50-90% of pregnant women and is often dismissed as a normal part of pregnancy. However, the long-term consequences can be dramatic. Up to 21% of women with PLPP still have pain three years postpartum, and 10% experience disability, poorer quality of life, and lower ability to work 11 years after delivery. Because the multifactorial etiology of PLPP is unclear, prevention and treatment fall short. Previous studies on the causes of PLPP focused on impairments in motor output but ignored that impairments in sensory input (e.g., proprioception, the primary expertise of our research group) often precede motor output problems. Moreover, though psychological factors such as fear (of movement) are known to affect PLPP, their predictive role in PLPP remains understudied. Finally, the role of systemic inflammation in PLPP has yet to be examined, despite recent studies demonstrating its role in the chronification of lumbopelvic pain in the general population.

This prospective cohort study aims to identify new modifiable predictors for the onset of PLPP during pregnancy and its persistence postpartum. The investigators will compare sensory (proprioception, body perception), fear-related, and inflammatory factors between women with and without PLPP and determine their predictive role in the onset and persistence of PLPP. The results will increase our understanding of the multifactorial etiology of PLPP and help optimize prevention and treatment.

DETAILED DESCRIPTION:
This study comprises a prospective cohort study with three objectives.

Objective 1 is to investigate whether the reliance on lumbar versus ankle proprioception during standing and body perception at the lower back (i.e., "proprioceptive factors"), anxiety, fear of movement, pain catastrophizing, depression, stress, and coping with stressful situations (i.e. "fear-related factors"), and inflammatory markers (i.e., "inflammatory factors") change over time and differ between women with and without PLPP in the 3rd pregnancy trimester, 6 weeks postpartum, and 9 months postpartum. We hypothesize that women with PLPP show (1a) a maladaptive reliance on ankle proprioception and/or disturbed body perception at the lower back, (1b) higher levels of fear of movement, anxiety, stress, depression, pain catastrophizing and poorer coping with stress, and (1c) greater immune activation and a disturbed balance of pro- vs. anti-inflammatory markers compared to pain-free women.

Objective 2 is to determine whether the proprioceptive, fear-related, and inflammatory factors are correlated in women with PLPP. Based on previous findings, we hypothesize that anxiety correlates with higher concentrations of IL-6 and IL-12, and lower concentrations of IL-2 and IL-10. We will also examine whether maladaptive reliance on ankle proprioception and disturbed body perception at the lower back correlate with fear of movement, anxiety, and concentrations of inflammatory markers in women with PLPP.

Objective 3 is to investigate whether the proprioceptive, fear-related, and inflammatory factors predict the presence of PLPP in the 3rd trimester, 6 weeks postpartum and 9 months postpartum. Based on previous research, we hypothesize that a maladaptive reliance on ankle proprioception and disturbed body perception at the lower back, higher levels of anxiety and fear of movement, and immune activation and disturbed balance of pro- and anti-inflammatory markers in the 1st trimester predict having PLPP in the 3rd trimester. We also expect that the presence of these factors in the 3rd trimester predicts the persistence of PLPP 6 weeks and 9 months postpartum.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent to participate
* 18-40 years old
* Pregnant
* Singleton pregnancy (confirmed through ultrasound)
* No current PLPP
* Dutch- or English-speaking

Exclusion Criteria:

* Pregnant for more than 16 weeks
* Currently experiencing PLPP, or having had PLPP during the index pregnancy
* History of surgery or major trauma to the spine or pelvis, major trauma or surgery to the lower limbs more than 2 years ago with current residual symptoms (e.g., pain, instability, stiffness), major trauma or surgery to the lower limbs less than 2 years ago
* Specific vestibular or balance disorders
* Use of medication that could affect balance (e.g., ototoxic or centrally-acting drugs)
* Having a medical diagnosis for, being treated by a rheumatologist for, or taking medication for a rheumatic condition
* (History of) a neurological disorder (e.g., neuropathy)
* Problems with vision that are not corrected by glasses, contact lenses or surgical eye correction
* Recent history of ankle problem (e.g., ankle sprain less than 3 weeks ago)
* Being on absolute/relative bed rest due to pregnancy complications
* (History of) inflammatory (e.g., gout, endometriosis), (auto)immune (e.g., lupus, ankylosis spondylitis, rheumatoid arthritis, psoriasis, Crohn's disease, Graves' disease, Hashimoto's thyroiditis, colitis ulcerosa, multiple sclerosis, etc.), hypothyroidism, or cancer.
* Having (had) a formal diagnosis of a psychiatric disorder (e.g., psychotic disorder).

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 211 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2028-09-01 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Pregnancy-related lumbopelvic pain (PLPP) (pregnant women) | Timepoint 2 (between gestational weeks 32-36), Timepoint 3 (6 weeks postpartum), Timepoint 4 (9 months postpartum)
  The presence of PLPP will be questioned at each timepoint. PLPP will be defined as: "self-reported pain in the lumbar area, between the twelfth rib and the gluteal fold, with or without pain between the posterior iliac crest and the gluteal fold, articularly in the vicinity of the sacroiliac joints, that may radiate to the posterior thigh and could occur separately or in conjunction with pain in the symphysis pubis."
Postural control (pregnant women) | Timepoint 1 (between gestational weeks 9-16), Timepoint 2 (between gestational weeks 32-36), Timepoint 3 (6 weeks postpartum), Timepoint 4 (9 months postpartum)
  Upright standing balance control will be measured as center-of-pressure displacements with a force plate.
Proprioceptive use during postural control (pregnant women) | Timepoint 1 (between gestational weeks 9-16), Timepoint 2 (between gestational weeks 32-36), Timepoint 3 (6 weeks postpartum), Timepoint 4 (9 months postpartum)
  Center-of-pressure displacements in response to ankle muscle and lower back muscle vibration (60 Hz, 15s) during upright standing will be measured with a force plate.
Inflammation with blood samples (pregnant women) | Timepoint 1 (between gestational weeks 9-16), Timepoint 2 (between gestational weeks 32-36), Timepoint 3 (6 weeks postpartum), Timepoint 4 (9 months postpartum)
  Serum concentrations of inflammatory mediators will be measured.
Task-related fear of movement (pregnant women) | Timepoint 1 (between gestational weeks 9-16), Timepoint 2 (between gestational weeks 32-36), Timepoint 3 (6 weeks postpartum), Timepoint 4 (9 months postpartum)
  Participants will be asked whether they are reluctant to perform any movement or activity in which their lower back or pelvis is involved, because they might have some concerns. If so, they are asked to specify the concerns and describe the movements or activities. For each of the activities, they will be asked to rate their (1) pain intensity, (2) perceived harmfulness, (3) fear, and (4) self-efficacy to perform the task, all via a Visual Analogue Scale (VAS) with 0= no pain/harmfulness/fear/self-efficacy to 100= maximal pain/harmfulness/fear/self-efficacy.
The ability to cope in a stressful situation with the Sense of Coherence Scale (SOC-13) (pregnant women) | Timepoint 1 (between gestational weeks 9-16), Timepoint 2 (between gestational weeks 32-36), Timepoint 3 (6 weeks postpartum), Timepoint 4 (9 months postpartum)
  The SOC-13 contains 13 items, total score ranges 0 - 91.
Depression, anxiety and stress in general with the Depression Anxiety Stress Scale (DASS-21) (pregnant women) | Timepoint 1 (between gestational weeks 9-16), Timepoint 2 (between gestational weeks 32-36), Timepoint 3 (6 weeks postpartum), Timepoint 4 (9 months postpartum)
  The DASS-21 evaluates depressive mood, anxiety and stress in general: 21 items, total score per subscale (Depression, Stress, Anxiety) range 0 - 21. Higher scores indicate higher levels of depressive mood (DASS-21-Depression), anxiety (DASS-21-Anxiety) and stress (DASS-21-Stress).
Pregnancy-related anxiety with the Revised Pregnancy-related Anxiety Questionnaire (PRAQ-R2) (pregnant women) | Timepoint 1 (between gestational weeks 9-16), Timepoint 2 (between gestational weeks 32-36)
  The PRAQ-R2 evaluates pregnancy-related anxiety: 10 items, total score range 10 - 50. Higher scores indicate higher levels of pregnancy-related anxiety.
Pregnancy-related depression with the Edinburgh Depression Scale (EDS)(pregnant women) | Timepoint 1 (between gestational weeks 9-16), Timepoint 2 (between gestational weeks 32-36), Timepoint 3 (6 weeks postpartum), Timepoint 4 (9 months postpartum)
  The EDS evaluates perinatal depression: 10 items, total score range 0 - 30. Higher scores indicate higher levels of pregnancy-related depression.
Catastrophic thinking related to pain with the Pain Catastrophizing Scale (PCS) (pregnant women) | Timepoint 1 (between gestational weeks 9-16), Timepoint 2 (between gestational weeks 32-36), Timepoint 3 (6 weeks postpartum), Timepoint 4 (9 months postpartum)
  The PCS contains 13 statements on thoughts and emotions possibly related to the experience of pain, for which the participants rates her agreement: 13 items, total score range 0 - 52. Higher scores indicate higher levels of pain catastrophizing.
Body perception at the lumbar spine assessed with a laterality recognition task ("Recognise Back" app) (pregnant women) | Timepoint 1 (between gestational weeks 9-16), Timepoint 2 (between gestational weeks 32-36), Timepoint 3 (6 weeks postpartum), Timepoint 4 (9 months postpartum)
  During the laterality recognition task, participants view 40 pictures of a model that has its lower back bent or rotated to the left or the right side. They will be asked to judge the direction of movement as quickly and accurately as possible. Average speed (in seconds) of response time and average accuracy of the answers (in %) will be recorded.
Body perception at the lumbar spine assessed with the Fremantle Back Awareness Questionnaire (FreBAQ) (pregnant women) | Timepoint 1 (between gestational weeks 9-16), Timepoint 2 (between gestational weeks 32-36), Timepoint 3 (6 weeks postpartum), Timepoint 4 (9 months postpartum)
  The FreBAQ assesses back-specific body perception: 9 items, total score range 0 - 45. Higher score indicate a more disturbed body perception.

SECONDARY OUTCOMES:
Disability due to PLPP with the Modified Oswestry Disability Index (mODI) (pregnant women) | Timepoint 1 (between gestational weeks 9-16), Timepoint 2 (between gestational weeks 32-36), Timepoint 3 (6 weeks postpartum), Timepoint 4 (9 months postpartum)
  The ODI is a 10-item self-report questionnaire that quantifies the extent of functional limitation in daily life due to low back pain. Each item is given a score between 0 (no limitation) and 5 (maximal limitation). The sum of the scores is multiplied by 2 to obtain a percentage score, with higher scores representing greater functional disability
Disability due to PLPP with the Quebec Back Pain Disability Scale (QBPDS) (pregnant women) | Timepoint 1 (between gestational weeks 9-16), Timepoint 2 (between gestational weeks 32-36), Timepoint 3 (6 weeks postpartum), Timepoint 4 (9 months postpartum)
  The QBPDS assesses disability in individuals with low back pain and PLPP: 20 items, total score range 0 - 100. Higher scores indicate higher levels of disability.
Pain intensity of PLPP with Visual Analogue Scale (VAS) (pregnant women) | Timepoint 2 (between gestational weeks 32-36), Timepoint 3 (6 weeks postpartum), Timepoint 4 (9 months postpartum)
  The participants will be asked to rate the pain intensity at the lower back or pelvic girdle they experience at this moment (i.e., both at the start and the end of the full test procedure), the average pain intensity during the past week, the minimal pain intensity during the past week, and the maximal pain intensity during the past week, by using the Visual Analogue Scale (VAS, 0-100), with 0 = "no pain" and 100 = "the worst pain imaginable".
Pain frequency of PLPP (pregnant women) | Timepoint 2 (between gestational weeks 32-36), Timepoint 3 (6 weeks postpartum), Timepoint 4 (9 months postpartum)
  The participants will be asked how often they experience pain (1= some days, 2= most days, 3= every day)
Health-related quality of life with the 36-Item Short Form Health Survey (SF-36) (pregnant women) | Timepoint 1 (between gestational weeks 9-16), Timepoint 2 (between gestational weeks 32-36), Timepoint 3 (6 weeks postpartum), Timepoint 4 (9 months postpartum)
  The SF-36 evaluates health-related quality of life, 8 scales: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health. Scores for the different scales are converted and pooled using a scoring key, for a total score ranging 0 - 100
Fear avoidance beliefs with the Fear-Avoidance Beliefs Questionnaire (FABQ) (pregnant women) | Timepoint 1 (between gestational weeks 9-16), Timepoint 2 (between gestational weeks 32-36), Timepoint 3 (6 weeks postpartum), Timepoint 4 (9 months postpartum)
  The FABQ consists of 16 statements for which the participant rates her agreement with the statement on a scale from 0 ("completely disagree") to 6 ("completely agree"): 16 items, total score range 0 - 96). Higher scores on the FABQ indicated more strongly held fear-avoidance beliefs.
Pain location of PLPP with a body chart (pregnant women) | Timepoint 2 (between gestational weeks 32-36), Timepoint 3 (6 weeks postpartum), Timepoint 4 (9 months postpartum)
  Individuals with PLPP will indicate the pain locations on a body chart.
Current body weight (pregnant women) | Timepoint 1 (between gestational weeks 9-16), Timepoint 2 (between gestational weeks 32-36), Timepoint 3 (6 weeks postpartum), Timepoint 4 (9 months postpartum)
  Current body weight will be measured (kg)
Current fat mass (in kg) and fat-free mass (in kg) (pregnant women) | Timepoint 1 (between gestational weeks 9-16), Timepoint 2 (between gestational weeks 32-36), Timepoint 3 (6 weeks postpartum), and Timepoint 4 (9 months postpartum)
  Current fat mass and fat-free mass (in kg) will be measured using bioelectrical impedance analysis (Bodystat 1500, EuroMedix).
Current total body water (in liter) (pregnant women) | Timepoint 1 (between gestational weeks 9-16), Timepoint 2 (between gestational weeks 32-36), Timepoint 3 (6 weeks postpartum), and Timepoint 4 (9 months postpartum)
  Current total body water (in liter) will be measured using bioelectrical impedance analysis (Bodystat 1500, EuroMedix).

OTHER OUTCOMES:
Diagnostic clinical tests for PLPP (pregnant women) | Timepoint 2 (between gestational weeks 32-36), Timepoint 3 (6 weeks postpartum), Timepoint 4 (9 months postpartum)
  In case the participant indicates pain in (one of) the PLPP regions (first criterium), the following clinical tests will be performed (second criterium) to confirm the presence of PLPP: thigh thrust, modified Trendelenburg test, Active straight leg raise test (ASLR).
  The participant will perform the ASLR test in supine lying: she will be asked to lift one leg 20 cm off the bed, and a score between 0 and 5 will be assigned depending on the difficulty experienced (0= "not difficult at all, 1= minimally difficult, 2= somewhat difficult, 3 = fairly difficult, 4= very difficult, 5= unable to do).
Sociodemographic information: age (pregnant women) | Timepoint 1 (between gestational weeks 9-16)
  The age of the participant will be noted (in years and months)
Sociodemographic information: annual household income (pregnant women) | Timepoint 1 (between gestational weeks 9-16)
  The participant will be asked: How would you describe your ability to make ends meet, considering your income and expenses?: With great difficulty, with difficulty, with some difficulty, fairly easily, easily, very easily
Sociodemographic information: marital status (pregnant women) | Timepoint 1 (between gestational weeks 9-16)
  Marital status will be questioned (having a partner or not, living together/alone)
Sociodemographic information: educational level (pregnant women) | Timepoint 1 (between gestational weeks 9-16)
  Highest obtained educational level will be recorded (i.e., primary education, secondary education, higher education (e.g., bachelor, master, PhD), currently in secondary education, currently in higher education)
Sociodemographic information: current employment status (pregnant women) | Timepoint 1 (between gestational weeks 9-16), Timepoint 2 (between gestational weeks 32-36), Timepoint 3 (6 weeks postpartum), Timepoint 4 (9 months postpartum)
  Current job status will be recorded (i.e., paid full-time job, paid part-time job, in sick leave because of issues related to pregnancy but not due to PLPP, in sick leave because of PLPP, in sick leave for reasons not related to pregnancy or PLPP, paid job but currently on career break (e.g., pregnancy or maternity leave), unemployed, no paid job but unpaid volunteer work, student), and type of work (i.e., sedentary, manual work, heavy manual work)
Number of previous miscarriages (pregnant women) | Timepoint 1 (between gestational weeks 9-16)
  The number of previous miscarriages will be recorded.
Smoking habits (pregnant women) | Timepoint 1 (between gestational weeks 9-16), Timepoint 2 (between gestational weeks 32-36), Timepoint 3 (6 weeks postpartum), Timepoint 4 (9 months postpartum)
  Smoking habits, including tobacco and vaping (i.e., daily, occasional, former, non-smoker) and number of cigarettes per day will be questioned.
Alcohol consumption (pregnant women) | Timepoint 1 (between gestational weeks 9-16), Timepoint 2 (between gestational weeks 32-36), Timepoint 3 (6 weeks postpartum), Timepoint 4 (9 months postpartum)
  Alcohol consumption (i.e., lifetime abstainer, former infrequent drinker, former regular drinker, current infrequent drinker, current light drinker, current moderate drinker, current heavier drinker) will be questioned.
Physical activity with IPAQ-SF (pregnant women) | Timepoint 1 (between gestational weeks 9-16), Timepoint 2 (between gestational weeks 32-36), Timepoint 3 (6 weeks postpartum), Timepoint 4 (9 months postpartum)
  Score on the International Physical Activity Questionnaire short form (IPAQ-SF).
Pain location apart from PLPP with a body chart (pregnant women) | Timepoint 1 (between gestational weeks 9-16), Timepoint 2 (between gestational weeks 32-36), Timepoint 3 (6 weeks postpartum), Timepoint 4 (9 months postpartum)
  All women will be asked whether they experience any recurrent or continuous pain apart from PLPP, and to indicate the pain locations on a body chart.
Subjective sleep quality with the Pittsburgh Sleep Quality Index (PSQI) (pregnant women) | Timepoint 1 (between gestational weeks 9-16), Timepoint 2 (between gestational weeks 32-36), Timepoint 3 (6 weeks postpartum), Timepoint 4 (9 months postpartum)
  The PSQI assesses sleep quality over the past month: 19 items, global sleep quality scores range 0 - 21.
Height (pregnant women) | Timepoint 1 (between gestational weeks 9-16)
  Height will be measured and reported in cm.
Pre-pregnancy body weight (pregnant women) | Timepoint 1 (between gestational weeks 9-16)
  Pre-pregnancy body weight will be questioned and reported in kg.
Falls during current pregnancy or in postpartum period (pregnant women) | Timepoint 1 (between gestational weeks 9-16), Timepoint 2 (between gestational weeks 32-36), Timepoint 3 (6 weeks postpartum), Timepoint 4 (9 months postpartum)
  The investigators will ask the participants whether they have sustained any falls during their current pregnancy (number of falls, gestational week during which fall(s) occurred, situation during which fall occurred (trip, slip, during stair ascent, during stair descent, during athletic activity), and injury severity associated with fall (no injury, mild injury requiring home treatment, major injury requiring medical attention))
Pelvic floor symptoms with the PFDI-20 (pregnant women) | Timepoint 1 (between gestational weeks 9-16), Timepoint 2 (between gestational weeks 32-36), Timepoint 3 (6 weeks postpartum), Timepoint 4 (9 months postpartum)
  Pelvic floor symptoms, i.e., urinary incontinence, fecal incontinence and pelvic organ prolapse will be assessed with the validated 20-item Pelvic Floor Distress Inventory (PFDI-20). The PFDI-20 contains 20 items, total score range 0 - 300.
Workload (pregnant women) | Timepoint 1 (between gestational weeks 9-16), Timepoint 2 (between gestational weeks 32-36), Timepoint 3 (6 weeks postpartum), Timepoint 4 (9 months postpartum)
  The participants will be asked whether they worked in uncomfortable positions, performed irregular work, or did shifts during pregnancy and postpartum.
Low back pain, pelvic girdle pain and pain conditions (pregnant women) | Timepoint 1 (between gestational weeks 9-16)
  The participants will be asked if they have a history of low back pain, pelvic girdle pain or other (chronic) pain conditions.
Previous stillbirths and live births | Timepoint 1 (between gestational weeks 9-16)
  The number of previous stillbirths and live births will be recorded.
Number of falls during previous pregnancies | Timepoint 1 (between gestational weeks 9-16)
  The investigators will ask the participants whether they have sustained any falls during their previous pregnancy (number of falls, situation during which fall occurred (trip, slip, during stair ascent, during stair descent, during athletic activity), and injury severity associated with fall (no injury, mild injury requiring home treatment, major injury requiring medical attention))
Urinary and anal incontinence during previous pregnancies (pregnant women) | Timepoint 1 (between gestational weeks 9-16)
  The presence of urinary and anal incontinence during previous pregnancies (yes/no), and the recovery postpartum (full, partial, no recovery) will be questioned.
Information on previous deliveries (pregnant women) | Timepoint 1 (between gestational weeks 9-16)
  For each of the previous deliveries, we will ask birth weight, maternal age at time of delivery, delivery mode (vaginal, c-section), instrumented delivery (no, forceps extraction, vacuum extraction, fundal pressure), whether the delivery was induced (yes, no), whether a vaginal tear or episiotomy was present (episiotomy, tear, no), and whether the pregnancy was through assisted reproductive treatment (yes, no).
History of PLPP during previous pregnancies | Timepoint 1 (between gestational weeks 9-16)
  All participants will be asked whether they experienced PLPP during previous pregnancies (yes,no), and if yes, the total duration in weeks, the pain frequency (1= some days, 2= most days, 3= every day), whether they experienced one episode of PLPP or whether PLPP was recurrent or continuous, whether PLPP persisted postpartum and for how many weeks, and whether they sought medical help for PLPP and/or whether the pain was disabling or whether they required sick leave.

CONTACTS AND LOCATIONS:
Overall Officials: Lotte Janssens, Prof, PhD, PT, Principal Investigator — Hasselt University; Inge Geraerts, Prof, PhD, PT, Principal Investigator — KU Leuven
Locations (2):
- Belgium (2):
  - Hasselt University, Hasselt
  - KU Leuven, Leuven

IPD SHARING:
Plan to Share IPD: No